CLINICAL TRIAL: NCT01949142
Title: Prospective, Randomized, Double-Blind, Sham-Controlled, Multicenter, P3 Study of OTO-201 Given as a Single IT Injection For Intra-Operative Treatment of Middle Ear Effusion in Pediatric Subjects Requiring Tympanostomy Tube Placement
Brief Title: OTO-201 for the Treatment of Middle Ear Effusion in Pediatric Subjects Requiring Tympanostomy Tube Placement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otonomy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201-201302
Record Dates: First submitted 2013-09-20; First posted 2013-09-24 (Estimated); Results first posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-05

CONDITIONS: Otitis Media With Effusion
Keywords: otitis media; otorrhea; middle ear effusion; tympanostomy tubes
MeSH Terms: conditions — Otitis Media with Effusion; Otitis Media | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OTO-201 (Experimental): OTO-201: Single, intratympanic injection:
  One injection of 6 mg OTO-201 (ciprofloxacin in poloxamer 407) into each ear during surgery.
  Interventions: Drug: OTO-201
- Sham (Sham Comparator): Sham: Simulated single, intratympanic injection:
  One sham injection into each ear during surgery.
  Interventions: Drug: Sham

INTERVENTIONS:
Drug: OTO-201 — Single, intratympanic injection
  Arms: OTO-201
Drug: Sham — Simulated single, intratympanic injection
  Arms: Sham

SUMMARY:
The purpose of this study is to confirm the effectiveness, safety and tolerability of OTO-201 in the treatment of pediatric subjects with bilateral middle ear effusion who require tympanostomy tube placement.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, sham-controlled, multicenter, Phase 3 study of OTO-201 administered intraoperatively in pediatric subjects with bilateral middle ear effusion requiring TT (tympanostomy tube) placement. One dose level (6 mg) of OTO-201 was evaluated relative to sham (empty syringe).

Study subjects are required to have a clinical diagnosis of bilateral middle ear effusion requiring TT placement. On the day of surgery, prior to surgery, eligible subjects were examined via otoscope to confirm bilateral middle ear effusion. Subjects with bilateral middle ear effusion were randomized to either 6 mg OTO-201 or sham. Subjects without bilateral effusion on the day of surgery were not randomized and were considered screen failures.

Approximately 264 subjects are planned to be randomized to OTO-201 or sham using a 2:1 allocation ratio. Randomization to OTO-201 or sham was stratified by age: 6 months to 2 years or >2 years.

Subjects are to visit the study site for safety assessments and otoscopic examination on Days 4, 8, 15, and 29. The assessment of otorrhea by the blinded assessor for the primary efficacy endpoint occurred on Days 4, 8, and 15.

ELIGIBILITY:
Inclusion Criteria includes, but is not limited to:

* Subject is a male or female aged 6 months to 17 years, inclusive
* Subject has a clinical diagnosis of bilateral middle ear effusion requiring tympanostomy tube placement
* Subject's caregiver is willing to comply with the protocol and attend all study visits

Exclusion Criteria includes, but is not limited to:

* Subject has a history of prior ear or mastoid surgery, not including myringotomy or myringotomy with tympanostomy tube placement
* Subject has a history of sensorineural hearing loss
* Subject has a history of chronic or recurrent bacterial infections other than otitis media that likely will require treatment with antibiotics during the course of the study

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 266 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl LeBel, PhD, Study Director — Otonomy, Inc.
Locations (1):
- Call/email Otonomy Central Contact for Trial Locations, San Diego, California, United States

REFERENCES:
- [Derived] Mair EA, Park AH, Don D, Koempel J, Bear M, LeBel C. Safety and Efficacy of Intratympanic Ciprofloxacin Otic Suspension in Children With Middle Ear Effusion Undergoing Tympanostomy Tube Placement: Two Randomized Clinical Trials. JAMA Otolaryngol Head Neck Surg. 2016 May 1;142(5):444-51. doi: 10.1001/jamaoto.2016.0001. PMID 26985629

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 29 centers, 25 in the United States and 4 from Canada.
Pre-assignment Details: The reporting group includes all randomized participants (n=266)
Period: Overall Study
Arm/Group | OTO-201 | Sham
Started | 179 | 87
Completed | 176 | 86
Not Completed | 3 | 1
Not completed — Withdrawal of consent | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Parent changed their mind | 1 | 0

BASELINE CHARACTERISTICS:
Population: The reporting group includes all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | OTO-201 | Sham | Total
Number analyzed (Participants) | 179 | 87 | 266
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.392 (2.0710) | 2.463 (2.1176) | 2.416 (2.0826)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 31 | 106
  Male | 104 | 56 | 160

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Treatment Failures
Description: Cumulative proportion of treatment failures:
  The efficacy endpoint for both trials was the cumulative proportion of study treatment failures through Day 15, defined as the occurrence of any of the following events: otorrhea as determined by a blinded assessor on or after 3 days post-surgery, otic or systemic antibacterial drug use for any reason any time post-surgery, as well as patients who missed visits or were lost-to-follow-up.
Time Frame: Day 15 - 2 weeks after dosing
Population: Full Analysis Set
Measure: Number; unit: percentage of treatment failures
Arm/Group | OTO-201 | Sham
Number analyzed (Participants) | 179 | 87
percentage of treatment failures | 24.6 | 44.8

2. Secondary Outcome: Evaluation of Adverse Events, Otoscopic Exams, Audiometry, and Tympanometry
Description: Safety variables included the frequency of adverse events (AEs) and results from otoscopic examinations, tympanometry, audiometry, vital sign measurements, and physical examinations.
Time Frame: Up to one month
Population: Safety Analysis Set (number of ears is equivalent to number of participants)
Measure: Number; unit: percentage of ears
Arm/Group | OTO-201 | Sham
Number analyzed (Participants) | 179 | 86
percentage of ears
  Otoscopic abnormal exams @ day 29-left ear | 1.1 | 2.4
  Otoscopic abnormal exams @ day 29-right ear | 0.6 | 0.0
  Audiometry Patent tubes @ day 29-left ear | 98.3 | 94.1
  Audiometry Patent tubes @ day 29-right ear | 96.0 | 96.5
  Tympanometry Category of B (large) day 29-left ear | 89.2 | 84.1
  Tympanometry Category of B (large)day 29-right ear | 91.0 | 88.9

3. Secondary Outcome: Microbiological Response
Description: Subjects whose samples tested positive for bacteria in either or both ears.
Time Frame: Day 15 - 2 weeks after dosing
Population: Microbiologically Evaluable Set
Measure: Number; unit: percentage of Microbiological response
Arm/Group | OTO-201 | Sham
Number analyzed (Participants) | 41 | 22
percentage of Microbiological response | 81 | 41

ADVERSE EVENTS:
Time Frame: Up to 6 weeks for each subject with total study time of 7 months. All AEs reported or observed after the informed consent had been signed and during or after dosing with the study drug were recorded on the AE page of the eCRF for all randomized subjects.
Groups:
- OTO-201 Single, Intratympanic Injection: OTO-201: One injection of 6 mg OTO-201 (ciprofloxacin in poloxamer 407) into each ear during surgery.
- Sham-Simulated Single, Intratympanic Injection: Sham: One sham injection into each ear during surgery.
Arm/Group | OTO-201 Single, Intratympanic Injection | Sham-Simulated Single, Intratympanic Injection
Serious Adverse Events (participants affected / at risk) | 3/179 | 0/86
Other Adverse Events (participants affected / at risk) | 64/179 | 28/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTO-201 Single, Intratympanic Injection (N=179) | Sham-Simulated Single, Intratympanic Injection (N=86)
Bronchiolitis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OTO-201 Single, Intratympanic Injection (N=179) | Sham-Simulated Single, Intratympanic Injection (N=86)
Irritability (General disorders) | 10 | 2
Nasopharyngitis (Infections and infestations) | 12 | 4
Upper respiratory tract infection (Infections and infestations) | 11 | 3
Teething (Gastrointestinal disorders) | 11 | 3
Pyrexia (General disorders) | 15 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
From the Protocol:

14.11. Use of Information and Publication. All information concerning OTO-201...remains the sole property of Otonomy. Any publication or other public presentation of results from this study requires prior review and written approval of Otonomy. Draft abstracts, manuscripts, and materials for presentation at scientific meetings should be provided to the sponsor at least 30 working days prior to abstract or other relevant submission deadlines.